CLINICAL TRIAL: NCT00658047
Title: A Phase II, Multi-center, Randomized, Double-blind, Methotrexate Controlled Study to Assess the Clinical Efficacy, Safety, and Tolerability of CH-1504 in Subjects With Active Rheumatoid Arthritis
Brief Title: A Study to Assess CH1504 in Patients With Active Rheumatoid Arthritis
Acronym: CH-1504-201
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chelsea Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CH-1504-201
Record Dates: First submitted 2008-04-08; First posted 2008-04-14 (Estimated); Last update posted 2013-04-15 (Estimated); Status verified 2013-04

CONDITIONS: Arthritis, Rheumatoid
Keywords: Arthritis, Rheumatoid; Phase II; Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — 4'-methylene-5,8,10-trideazaaminopterin; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 0.25 mg CH-1504 (Experimental): 0.25 mg CH-1504
  Interventions: Drug: CH-1504
- 0.5 mg CH-1504 (Experimental): 0.5 mg CH-1504
  Interventions: Drug: CH-1504
- 1.0 mg CH-1504 (Experimental): 1.0 mg CH-1504
  Interventions: Drug: CH-1504
- Methotrexate (Active Comparator): Methotrexate (MTX) 10 mg/week for 2 weeks, 15 mg/week for 2 weeks, 20 mg/week for 8 weeks
  Interventions: Drug: Methotrexate (MTX)

INTERVENTIONS:
Drug: CH-1504 — Comparison of different doses of CH-1504
  Arms: 0.25 mg CH-1504; 0.5 mg CH-1504; 1.0 mg CH-1504
Drug: Methotrexate (MTX) — 10mg/week for 2 weeks escalated to 15mg/week for 2 weeks escalated to 20mg/week for 8 weeks
  Other Names: amethopterin (previous name for MTX)
  Arms: Methotrexate

SUMMARY:
The purpose of this trial is to assess the clinical effect of CH-1504 at doses of 0.25, 0.5 and 1.0 mg per day in patients with active rheumatoid arthritis by determining the proportion of patients achieving an American College of Rheumatology (ACR) 20% improvement response.

DETAILED DESCRIPTION:
Rheumatoid Arthritis (RA) is a chronic inflammatory disease of unknown cause that leads to pain, stiffness, swelling and limitation of joint function. If left untreated, RA produces serious destruction of joints that frequently leads to permanent disability.

Methotrexate (MTX) is currently the most commonly prescribed first-line disease modifying anti-rheumatic drug (DMARD) because of its early onset of action, good efficacy, and ease of administration. In addition, MTX can be combined with other FDA approved DMARDs, including gold compounds, sulfasalazine, hydroxychloroquine, TNF inhibitors, anakinra and leflunomide. However, the administration of MTX has been associated with serious side effects such as skin reactions, pneumonitis, gastrointestinal disturbances including diarrhea, ulcerative stomatitis and hemorrhagic enteritis, hepatotoxicity and renal toxicity. Overall it is estimated that up to 30% of all patients discontinue MTX therapy due to side effects.

MTX enters cells via the Reduced Folate Carrier (RFC) system. Once inside cells, it is converted enzymatically to polyglutamylated derivatives. These metabolites cannot be readily effluxed and are retained in tissues. The accumulation of polyglutamyl metabolites of MTX for prolonged periods may play a significant role in both the efficacy and the toxicity of this compound. Methotrexate in its parent form only has activity against dihydrofolate reductase (DHFR). In order for it to have significant activity against other enzymes (i.e. Thymidylate Synthase (TS)) it must be polyglutamylated. However by being polyglutamylated the MTX metabolite is retained in the cell and may potentiate the cytotoxicity of MTX. In addition to polyglutamylation metabolism, MTX is also hydroxylated in the liver to a metabolite known as 7-hydroxymethotrexate, which is also subject to polyglutamylation and cell retention. This metabolite has been implicated in liver and kidney toxicity of the parent compound, while contributing no role in efficacy.

CH-1504 has been shown in vitro to be a nonpolyglutamylatable and nonhydroxylatable antifolate that is more efficiently taken up into cells by the reduced folate carrier (RFC) system than is MTX. CH-1504 has significant activity on both DHFR and TS enzymes without the need for polyglutamylation. The lack of hydroxylation potentially leads to enhanced levels of the active drug in the cell. Furthermore, the glutamyl moiety is not susceptible to being cleaved by carboxypeptidase. Thus CH-1504 may be referred to as a metabolically stable antifolate. It is our hypothesis that in the clinical setting CH-1504 will demonstrate the efficacy of classical antifolates (via folate enzyme inhibition) but will be devoid of the toxicity secondary to the formation of the polyglutamylated and hydroxylated metabolites, providing a significantly improved therapeutic index compared to classical antifolates, such as MTX.

This study is a randomized, double-blind, methotrexate controlled study to assess the clinical effect of CH-1504 in patients with active rheumatoid arthritis by determining the proportion of patients achieving an ACR20 response after 12 weeks of treatment.

Secondary objectives are:

* Assess the clinical efficacy of CH-1504 by proportion of patients achieving ACR50 and ACR70 responses.
* Assess the clinical efficacy of CH-1504 using EULAR "good" and "moderate" response criteria.
* Assess the clinical efficacy of CH-1504 using the difference from baseline of ACR core set and DAS28 of measures.
* Evaluate the safety and tolerability of CH-1504 in RA patients as determined by the frequency and severity of adverse events, laboratory abnormalities, and dropouts.
* Identify the dose response relationship of CH-1504

ELIGIBILITY:
Inclusion; To be eligible for inclusion, each patient must fulfill the following criteria:

* Patients must be between the ages of 18 and 80;
* Have been diagnosed with active rheumatoid arthritis according to ACR criteria;
* Have at least 6 swollen joints (max = 66) and 6 tender joints (max = 68) at screening and baseline visits;
* Patients must have at least one of the following:
* C-reactive protein > 1.0 mg/dl at screening;
* erythrocyte sedimentation rate > 20 mm/Hr;
* Morning stiffness > 45 min. at screening;
* Patients must have blood test values per the following criteria:
* ALT, AST < 1.2 U/l x ULN
* Albumin > 2.5 g/dl
* Prothrombin Time < 1.2 INR
* Hb > 9.0 g/dl
* Hct > 35%
* WBC > 3000 μl (mm3)
* Neutrophils > 1000 μl (mm3)
* Platelets > 100000 μl
* Creatinine < 1.2 mg/dl
* Patients must have voluntarily signed the informed consent

Exclusion; Patients are not eligible for this study if they fulfill one or more of the following criteria:

* Patients who received previous methotrexate therapy;
* Patients who received previous therapy with any biologic agent;
* Previous biologic therapy for a disease other than RA is permitted so long as their last dose was more than 120 days prior to baseline;
* Patients currently taking sulfasalazine;
* Previous sulfasalazine therapy is permitted so long as their last dose was more than 30 days prior to baseline;
* Patients currently taking hydroxychloroquine;
* Previous hydroxychloroquine is permitted so long as their last dose was more than 120 days prior to baseline;
* Female patients of child bearing potential who are pregnant or who are not using two methods of contraception (at least one barrier: i.e. condom) with their partner;
* Male patients who are sexually active and not using two methods of contraception (at least one barrier: i.e. condom) with their partner;
* Patients with any current active infection or infections requiring IV drug therapy within 30 days of baseline or oral therapy within 15 days of Baseline;
* Patients that have had any surgical procedures within 30 days of baseline;
* Patients with a history of HIV, Hepatitis B or C;
* Patients who consume more than 7 units of alcohol per week (1 unit = 5 ounces/150 ml of wine = 1.5 ounces/45 ml spirits = 12 ounces/360 ml of beer);
* Patients currently receiving any investigational drug or have received an investigational drug within 30 days of baseline or 5 half-lives of the investigational drug (whichever is longer);
* Patients with a history of cancer within the past 5 years other than a successfully treated, non-metastatic cutaneous squamous cell or basal cell carcinoma or cervical cancer in situ;
* Patients with a history of, or any, disease associated with an inflammatory arthritis other than RA;
* Patients with a chest X-ray that indicates the presence of pulmonary fibrosis (Chest x-ray may be taken with in 28 days of screening);
* Patients receiving Probenecid;
* Patients who have received any steroid injections within 30 days of baseline;
* Patients with concomitant diseases that are unstable (i.e. cardiac, pulmonary) or that may affect drug activity (i.e. absorption, reactions, change in kinetics);
* Patients considered by the investigator to be an unsuitable candidate to receive CH-1504;
* Wheelchair or bed-bound patients.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2008-04; Primary Completion 2009-02 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Assess the clinical effect of CH-1504 (0.25, 0.5, and 1.0 mg po daily) by determining the proportion of patients achieving an ACR20 response. | 3 months of treatment

SECONDARY OUTCOMES:
Assess the clinical efficacy of CH-1504 by proportion of patients achieving ACR50 and ACR70 responses. | 3 months of treatment
Assess the clinical efficacy of CH-1504 using EULAR "good" and "moderate" response criteria. | 3 months of treatment
Assess the clinical efficacy of CH-1504 using the difference from baseline of ACR core set and DAS28 of measures. | 3 months of treatment
Evaluate the safety and tolerability of CH-1504 in RA patients as determined by the frequency and severity of adverse events, laboratory abnormalities, and dropouts. | 3 months of treatment
Identify the dose response relationship of CH-1504. | 3 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Edward Keystone, MD, Principal Investigator — The Rebecca MacDonald Centre for Arthritis and Autoimmune Disease
Locations (1):
- The Rebecca MacDonald Centre for Arthritis and Autoimmune Disease, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Keystone EC, Shirinsky VS, Simon LS, Pedder S, Hewitt LA; CH-1504 Study Group. Efficacy and safety of CH-1504, a metabolically stable antifolate, in patients with active rheumatoid arthritis: results of a phase II multicenter randomized study. J Rheumatol. 2011 Sep;38(9):1875-83. doi: 10.3899/jrheum.101038. Epub 2011 Jul 1. PMID 21724705